CLINICAL TRIAL: NCT06820749
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of HSK31858 Tablets in Patients with Airway Mucus Hypersecretion in Chronic Airway Inflammatory Diseases
Brief Title: A Study to Evaluate the Efficacy and Safety of HSK31858 Tablets in Patients with Airway Mucus Hypersecretion
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31858-204
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Asthma Bronchiale; Bronchiectasis; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HSK31858 20mg (Experimental): multiple oral doses: 20mg/d for 12w
  Interventions: Drug: HSK31858
- HSK31858 40mg (Experimental): multiple oral doses: 40mg/d for 12w
  Interventions: Drug: HSK31858
- placebo (Placebo Comparator): multiple oral doses for 12w
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK31858 — HSK31858 is a novel inhibitor of DPP1 developed by Hisco Pharmaceutical and can reduce pulmonary exacerbations over a 12-week treatment period in patients with airway mucus hypersecretion in chronic airway inflammatory diseases
  Arms: HSK31858 20mg; HSK31858 40mg
Drug: Placebo — the placebo comparator of study
  Arms: placebo

SUMMARY:
This is a phase II, randomised, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of HSK31858 in patients with airway mucus hypersecretion in chronic airway inflammatory diseases

ELIGIBILITY:
Inclusion Criteria:

1)Able to fully understand and voluntarily sign informed consent; 2)Male or female patients ≥18 years of age at the time of screening; 3)Patient with chronic airway inflammatory diseases (bronchiectasis, chronic obstructive pulmonary disease, asthma); 4)24h sputum volume ≥10ml at screening period (V1) and baseline (V2); 5) If the subjects have used background therapy drugs, other background therapy drugs other than expectorant drugs were used to maintain stability for ≥1 month before screening; 6)Female subjects with fertility or male subjects whose partner is a female with fertility must agree to have no plans to have children and to use contraception voluntarily from the time of signing the informed consent form until 3 months after the last dose. All females of childbearing potential must have a negative screening pregnancy test.

7)Subjects are able to communicate well with the investigator and are able to complete the study in accordance with the protocol requirements.

Exclusion Criteria:

1. Known allergic history to the active ingredient of the investigational drug or other drugs with similar chemical structure;
2. FEV1 accounted for less than 30% of the estimated value after bronchodilator use;
3. Patients who have experienced any degree of acute exacerbation of asthma or are experiencing an acute exacerbation of asthma within 4 weeks prior to screening;
4. Hemoptysis (other than a small amount of bloody sputum or a blood clot smaller than a fingernail) occurs within 4 weeks prior to screening and requires urgent medical intervention;
5. Active infection or acute infection requiring systemic anti-infective therapy within 4 weeks prior to screening.
6. History of malignancy: subjects with basal cell carcinoma, limited squamous cell carcinoma of the skin, or cervical carcinoma in situ will be allowed to enter the study if curative treatment has been completed for at least 12 months prior to signing the informed consent form; subjects with other malignancies will be allowed to enter the study if curative treatment has been completed for at least 5 years prior to signing the informed consent form;
7. Presence of any severe and/or uncontrolled medical condition that, in the judgement of the investigator, affects the safety of the subject or interferes with the evaluation of the medication, including, but not limited to: severe neurological disease, history of serious mental disorders, major cardiovascular disease, diabetes mellitus that is poorly controlled on standardized therapy, presence of prolonged QTcF interval or cardiac arrhythmia, or immunodeficiency disorders;
8. Subjects with a history of liver disease or currently receiving treatment for liver disease during the screening period, including but not limited to acute and chronic hepatitis, cirrhosis or liver failure;
9. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg, and/or diastolic blood pressure ≥ 100 mmHg at screening or baseline);
10. Abnormal screening and baseline laboratory tests:

    1. White blood cell count < 3 × 109/L, or neutrophil count< 1.5 × 109/L, or platelet < 70 × 109/L, or hemoglobin < 90 g/L;
    2. Alanine aminotransferase (ALT) > 2 × ULN (upper limit of normal), or aspartate aminotransferase (AST) > 2 × ULN, or total bilirubin (TBIL) > 1.5 × ULN;
    3. Patients with moderate to severe renal insufficiency (eGFR < 60 ml/min/1.73m2, calculation of eGFR using the simplified MDRD equation);
11. Participation in a clinical trial of any other drug or medical device (treated with a drug or medical device in a clinical trial) within 1 months prior to screening;
12. Having received a drug that may cause hyperkeratosis of the skin (e.g., tumor necrosis factor alpha antagonist) within 4 weeks prior to screening;
13. Patients who have used a strong inducer or inhibitor of CYP3A within 14 days or 5 half-lives prior to the first investigational product administration, whichever is longer;
14. Comorbidities associated with the development of non-hereditary palmoplantar keratoderma (e.g., myxedema, chronic lymphoedema);
15. Comorbid periodontal disease that, in the judgement of the investigator, has an impact on the study;
16. Asthmatic currently smoking subjects or subjects who quit smoking within 6 months prior to the screening visit; previous smoking subjects with a smoking history >10 pack-year = packs per day × years of smoking (Note: 1 pack = 20 cigarettes, 10 pack-year = 1 pack/day × 10 years or 1/2 pack/day × 20 years).
17. History of drug use, or substance abuse within 2 years prior to screening;
18. Pregnant, or planning to become pregnant during the study, or breastfeeding;
19. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24 hour sputum weight | 12-week treatment period
  Change from baseline in 24 hour sputum weight after 12 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in expectoration difficulty score | 12-week treatment period
  Change from baseline in expectoration difficulty score after 4, 8 and 12 weeks of treatment.The expectoration difficulty score adopt a 4-level evaluation standard, 0 points for no expectoration, 1 points for easy expectoration, 2 points for moderate expectoration difficulty, and 3 points for hardest expectoration.
Change from baseline in sputum trait score | 12-week treatment period
  Change from baseline in sputum trait score after 4, 8, and 12 weeks of treatment.The sputum trait score was based on the Miller classification, according to the proportion of purulent part to total sputum volume.
Change from baseline in sputum viscosity score | 12-week treatment period
  Change from baseline in sputum viscosity score after 4, 8, and 12 weeks of treatment.The sputum viscosity score is based on a 5-level evaluation standard. Sputum adhering to the cup wall of the container and not sliding down is 1 point; sputum slowly sliding through the cup wall of the container under the action of gravity is 2 points; sputum sliding in large pieces through the cup wall under the action of gravity is 3 points; sputum is easily poured out and a small amount of thin mucus sticks to the cup wall of the container. No residual sputum on the wall of the container 5 points.
Change from baseline in cough severity score | 12-week treatment period
  Change from baseline in cough severity score after 4, 8, and 12 weeks of treatment.The visual analog scale (VAS) was used to score the severity of cough: a line 10 cm long was drawn on the white paper, and the corresponding scale was marked to indicate the severity of cough. The score was 0 to 10 points, 0 was no cough and no trouble to the patient, and 10 was the most serious cough and the most serious trouble to the patient.
Change from baseline in cough and sputum assessment questionnaire | 12-week treatment period
  Change from baseline in cough and sputum assessment questionnaire after 4, 8, and 12 weeks of treatment.The cough and sputum assessment questionnaire is an evaluation tool used to evaluate the impact of cough and sputum on the quality of life of patients. The contents involved four dimensions: cough symptoms, cough effects, sputum symptoms and sputum effects. Each dimension contained different items, which were scored and statistically converted, with a total score of 100 points. The lower the score, the heavier airway mucus hypersecretion.
Change from Baseline in forced expiratory volume in 1 second (FEV1) | 12-week treatment period
  Change from baseline in pre-bronchodilator forced expiratory volume in 1 second (FEV1) at 12 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality, China